CLINICAL TRIAL: NCT03615378
Title: A Randomized, Double Blind, Placebo Controlled Trial Evaluating Optimal Maintenance Strategies of Vitamin D Levels in Patients With Crohn's Disease in Remission
Brief Title: Maintenance Dosing of Vitamin D in Crohn's Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficulties with enrollment
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Gil Melmed, Clinical Director of Inflammatory Bowel Disease, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro50335
Record Dates: First submitted 2018-07-16; First posted 2018-08-03 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Crohns Disease; Vitamin D Deficiency
MeSH Terms: conditions — Crohn Disease; Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Vitamin D 1000 IU D3 daily (Active Comparator)
  Interventions: Dietary Supplement: 1000 IU D3
- Vitamin D 5000 IU D3 daily (Active Comparator)
  Interventions: Dietary Supplement: 5000 IU D3

INTERVENTIONS:
Dietary Supplement: 5000 IU D3 — Daily
  Arms: Vitamin D 5000 IU D3 daily
Dietary Supplement: 1000 IU D3 — Daily
  Arms: Vitamin D 1000 IU D3 daily
Dietary Supplement: Placebo — lactose/sugar tablet
  Arms: Placebo

SUMMARY:
Vitamin D repletion is important for bone health in patients with Crohn's disease. While repletion strategies in the general population yield similar results in those with Crohn's disease, maintenance strategies are variable. High quality evidence is lacking to determine the optimal strategy to maintain adequate levels of Vitamin D levels in patients with Crohn's disease.

DETAILED DESCRIPTION:
The investigators seek to identify patients with Crohn's disease in clinical remission who have vitamin D levels <30 ng/ml. Subjects will undergo a 8 week lead in period and receive Vitamin D supplementation with 50,000 IU D2 weekly for 8 weeks.Participants with sufficient Vitamin D levels after 8 weeks (>30 ng/mL) will be enrolled into the study and randomized to one of three arms: (1) placebo (2) 1000 IU/day Vitamin D3 (3) 5,000 IU/day Vitamin D3 for 22 weeks. Based on clinical experience, doses higher than the recommended doses for bone health in the general population (600-800 IU/day Vitamin D3) are needed to achieve and maintain optimal levels of Vitamin D in people with Crohn's disease.

The investigators aim to determine optimal maintenance dosing to sustain vitamin D sufficiency in people with Crohn's disease. The investigators also seek to determine demographic and disease related characteristics associated with inability to maintain sufficient levels.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Crohn's disease
2. In clinical remission as determined by the Harvey Bradshaw Index (CD) ≤4
3. 25(OH)D level <30 ng/ml within three months of study enrollment
4. Prior 25(OH)D level <30 ng/ml currently on repletion therapy
5. Provided written informed consent
6. 18 years of age or older
7. All maintenance therapies required to be on stable doses for 3 months.

Exclusion Criteria:

1. Unwilling to provide consent or lack capacity
2. Clinical disease activity (Harvey Bradshaw index >4)
3. Current pregnancy or attempting to conceive
4. Hypercalcemia (must have calcium level within 6 months of enrollment)
5. Known coexisting hyperparathyroidism
6. BMI >30 kg/m²
7. History of kidney stones
8. Subjects <18 years of age - pediatric population with different recommended dosing than adults
9. Non-english speakers
10. Has an ileo-anal pouch or ileostomy
11. C-reactive protein greater than 2x the upper limit of normal
12. Lactose intolerant
13. Short gut syndrome
14. Renal insufficiency (CrCl <60 ml/min)
15. Concomitant therapy with thiazide diuretics, barbiturates, digitalis or supplemental products containing vitamin D
16. Vitamin D levels <30ng/ml at completion of lead in

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Vitamin D serum level Vitamin D sufficiency | 22 weeks
  Serum level greater than or equal to 30 ng/ml

SECONDARY OUTCOMES:
Time to Vitamin D Insufficiency | 22 weeks
  Time (in weeks) from the measurement of sufficiency (at week 0) to Vitamin D insufficiency (defined as serum vitamin D level less than 30 ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: GIl Y Melmed, MD, MS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No information will be shared